CLINICAL TRIAL: NCT00161083
Title: Studie Naar De Effectiviteit Van Ursodeoxycholzuur Ter Preventie Van Galsteen-Gerelateerde Klachten Bij patiënten in Afwachting Van Een Cholecystectomie
Brief Title: UDCA for Symptomatic Gallstone Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dr. Falk Pharma GmbH (Industry); Dutch Digestive Diseases Foundation (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Agis Zorgverzekeringen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLDS WS 00-08; MLDS WS 00-08; ZonMw: 920-03-232
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2005-09

CONDITIONS: Cholecystolithiasis
Keywords: ursodeoxycholic acid; gallstone; complications; pancreatitis; gallbladder motility; colic
MeSH Terms: conditions — Cholecystolithiasis; Gallstones; Pancreatitis; Colic | interventions — Ursodeoxycholic Acid

INTERVENTIONS:
Drug: ursodeoxycholic acid

SUMMARY:
We conduct a randomized, double-blind, placebo-controlled trial on effects of UDCA on biliary pain and complications in highly symptomatic gallstone patients scheduled for cholecystectomy. We also evaluate potential beneficial effects of impaired gallbladder motility

DETAILED DESCRIPTION:
Gallstone disease is very common with an estimated prevalence of 10-15% in the adult Western population. Approximately 90% of gallstone carriers are asymptomatic. The annual risk of biliary colic in asymptomatic gallstone carriers has been suggested to be approximately 1%. Also, asymptomatic gallstone carriers are at risk for acute pancreatitis, choledocholithiasis and acute cholecystitis. Although accurate prospective data are lacking, annual incidences of these potentially lethal complications are estimated to be approximately 0.2%, 0.2% and 0.3%, respectively.

One can easily imagine that migration of gallbladder stones into the common bile duct may lead to biliary pain. How gallbladder stones remaining in the gallbladder lead to biliary symptoms is not entirely clear. Strong gallbladder contraction, with temporary impaction of the stone in the orifice of the cystic duct might cause biliary pain. Although impaired gallbladder motility could therefore theoretically protect against colics, symptomatic gallbladder stone patients often have complaints despite coexistent impaired gallbladder emptying.

Ursodeoxycholic acid (UDCA) has been claimed to reduce the risk of biliary pain, regardless of gallstone dissolution. In a large study by Tomida et al., risks of biliary pain or gallstone complications (acute cholecystitis) were reduced in both symptomatic and asymptomatic gallstone carriers, although gallstones were generally not dissolved. Also, biliary pancreatitis might be prevented by long-term UDCA treatment. Increased fasting and residual postprandial gallbladder volumes during UDCA treatment, less cholesterol crystals or decreased mucin contents in bile could be the underlying mechanisms for these beneficial effects. However, prospective studies on effects of UDCA on symptoms or complications in highly symptomatic patients are lacking.

In the Netherlands symptomatic gallstone patients are admitted to a waiting list for elective cholecystectomy by general surgeons. The waiting period may last several months because of logistic reasons. During this waiting period gallstone patients are at risk for biliary pain and complications. Therefore, we conducted a randomized, double-blind, placebo-controlled trial on effects of UDCA on biliary pain and complications in highly symptomatic gallstone patients scheduled for cholecystectomy. We also evaluated potential beneficial effects of impaired gallbladder motility

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age study are upon admission to the waiting list for elective cholecystectomy for symptomatic cholecystolithiasis defined as:

  * presence of gallbladder stones or sludge, without bile duct stones or bile duct dilatation at ultrasonography;\
  * at least one episode of severe right upper quadrant or midline epigastric pain of at least 30 min. duration, with radiation and/or movement urge, or at least three episodes of severe right upper quadrant or midline epigastric pain of at least 30 min. duration without such radiation or movement urge, in the previous 12 months

Exclusion Criteria:

* Contra-indication for general anaesthesia or surgery
* Current or previous acute cholecystitis, obstructive jaundice or pancreatitis
* Previous papillotomy, because of preferential flow of UDCA-enriched bile to the intestine rather than to the gallbladder
* Pregnancy or lactation
* Current or previous use of UDCA
* Participation in another study
* Inability to speak Dutch or English or mental disability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2001-11; Study Completion 2004-11

PRIMARY OUTCOMES:
incidence severe right upper quadrant or midline epigastric pain (> 30 min)and colic-free intervals

SECONDARY OUTCOMES:
nr gallstone complications (acute cholecystitis, choledocholithiasis or acute pancreatitis) and non-severe right upper quadrant or midline epigastric pain and nr aalgesics taken

CONTACTS AND LOCATIONS:
Overall Officials: Niels G Venneman, MD, Principal Investigator — UMC Utrecht; Karel J van Erpecum, MD, PhD, Study Director — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Venneman NG, Besselink MG, Keulemans YC, Vanberge-Henegouwen GP, Boermeester MA, Broeders IA, Go PM, van Erpecum KJ. Ursodeoxycholic acid exerts no beneficial effect in patients with symptomatic gallstones awaiting cholecystectomy. Hepatology. 2006 Jun;43(6):1276-83. doi: 10.1002/hep.21182. PMID 16729326